CLINICAL TRIAL: NCT04553744
Title: Survey of Extremity and Trunk Sarcoma Surgeons Regarding Surgical Management of Lymph Node Basins
Brief Title: Identification of Surgical Management of Lymph Node Basins and Surgical Practice Patterns Among Sarcoma Surgeons
Status: Withdrawn | Type: Observational
Why Stopped: 0 participant accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2020-0099; NCI-2020-06478 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0099 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-09-11; First posted 2020-09-17 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Soft Tissue Sarcoma; Lymph Node Cancer
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (survey): Participants complete an online survey over 5-10 minutes asking how they would manage lymph node basins in the extremity sarcoma.
  Interventions: Other: Survey Administration

INTERVENTIONS:
Other: Survey Administration — Complete survey

SUMMARY:
This study investigates the surgical management of lymph node basins for extremity and trunk soft tissue sarcoma (ETSTS) to identify and better understand the surgical practice patterns of sarcoma surgeons. ETSTS has been known to spread to distant locations including lymph nodes, with some subtypes of the disease spreading to lymph nodes more than others. This has led to sarcoma surgeons to treat patients differently from one another, including those with more lymph node involvement. The purpose of this study is to investigate the practice patterns of ETSTS surgeons.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Identify the practice patterns of sarcoma surgeons with respect to management of lymph node basins for extremity and trunk soft tissue sarcomas (ETSTS).

II. Identify when surgeons would perform sentinel lymph node biopsy and/or lymph node dissection for ETSTS and if management differs for high-risk subtypes of sarcoma that are more likely to have nodal metastases.

III. Identify differences in practice patterns between surgical oncologists and orthopedic oncologic surgeons.

OUTLINE:

Participants complete an online survey over 5-10 minutes asking how they would manage lymph node basins in the extremity sarcoma.

ELIGIBILITY:
Inclusion Criteria:

* Currently practicing surgeons who treat ETSTS and are members of The Society of Surgical Oncology and Musculoskeletal Tumor Society

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Practicing surgeons who are members of The Society of Surgical Oncology and Musculoskeletal Tumor Society, and treat extremity and trunk soft tissue sarcomas.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
Practice patterns of sarcoma surgeons | Up to 2 years
  Will identify the practice patterns of sarcoma surgeons with respect to management of lymph node basins for extremity and trunk soft tissue sarcomas (ETSTS).
Sentinel lymph node biopsy and/or lymph node dissection for ETSTS | Up to 2 years
  Will identify when surgeons would perform sentinel lymph node biopsy and/or lymph node dissection for ETSTS, and if management differs for high-risk subtypes of sarcoma that are more likely to have nodal metastases.
Differences in practice patterns | Up to 2 years
  Will identify differences in practice patterns between surgical oncologists and orthopedic oncologic surgeons.

CONTACTS AND LOCATIONS:
Overall Officials: Christina L Roland, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org